CLINICAL TRIAL: NCT07229833
Title: Validation of Fitbit Measurements in Hospitalized General Medicine Patients
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Robert Wu, Clinician Investigator, University Health Network, Toronto
Other Study IDs: 24-5399
Record Dates: First submitted 2025-07-29; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: GIM Diagnosis; Medicine; Admission to GIM
Keywords: wearable; sleep; heart rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- General internal medicine patients admitted to General Medicine Wards: Intervention: Fitbit Sense 2 (Fitbit, San Francisco, CA, USA)
  Gold standard devices: To compare measures, patients will be asked to wear the following for 24 hours:
  * Sleep study device - Nox T3 chest band with oximeter. Participants will be asked to wear this for 24 hours. The Nox T3 monitors chest movement and determines sleep stages. It is paired with a Nonin oximeter. This provides continuous oxygen saturation monitoring as well as heart rate and respiratory rate.
  * Step counter - An ankle-worn Stepwatch Activity Monitor which has been validated in hospital patients who move slowly.

SUMMARY:
Patients admitted to the General Internal Medicine ward are sick and in need of monitoring that cannot be provided at home or treatments best administered in hospital. Standard care currently includes vital signs measurements and in some cases ECG. Wearable devices that continuous monitor patients could provided added information to improve the care of inpatients. This could include more monitoring and catching deterioration before it happens. Wearables have been shown to be largely accurate for monitoring heart rate, however it is still necessary to determine if they can reliably measure sleep, activity, and other health metrics. For this, study investigators are evaluating the validity of FitBit Sense 2 (or other FitBit devices) for measurement of sleep, activity, heart rate, respiratory rate, and oxygen saturation.

ELIGIBILITY:
Subject inclusion criteria.

* General internal medicine patients admitted to General Medicine Wards.
* Able to consent.
* 18 years of age or older

Subject exclusion criteria.

* Patients who are purely palliative "comfort measures only" where measuring vital signs would not be appropriate and will be excluded.
* To reduce the potential risk of transmitting nosocomial infections, patients under contact precautions for methicillin resistant Staphylococcus aureus (MRSA) and Clostridium difficile infections will also be excluded.
* This study will also exclude patients at risk of vascular compromise of the arm or leg on which the wearable device was to be placed, such as patients with deep venous thrombosis, dialysis fistulas, and severe upper extremity trauma.
* Expected discharge less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be General Internal Medicine inpatients on the GIM wards. Patients who can provide informed consent will be approached for enrollment. Exclusion criteria are patients who are purely palliative and therefore in which vital sign measurement would be inappropriate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fitbit Sense 2 vs. StepWatch for activity (step count) | Collected over 24 hours in 1 min bins
  Comparisons of step counts between Fitbit and Modus StepWatch
Fitbit Sense 2 vs. Nox T3 for heart rate (bpm) | Fitbit collected over 24 hours in 1 min bins and Nox T3 collected during nighttime sleep in 1 sec bins
  Comparisons of HR between Fitbit and Nox pulse oximeter
Fitbit Sense 2 vs. Nox T3 for respiratory rate (breaths per minute) | Fitbit collected over 24 hours in 1 min bins and Nox T3 collected during nighttime sleep in 1 sec bins.
  Comparisons of RR between Fitbit and Nox RIP (respiratory inductive plethysmograph)
Fitbit Sense 2 vs. Nox T3 for oxygen saturation (SpO2, %) | Fitbit collected over 24 hours in 1 min bins and Nox collected during nighttime sleep in 1 sec bins.
  Comparisons of SpO2 between Fitbit and Nox T3
Fitbit Sense 2 vs. Nox T3 for total sleep time (min) | Fitbit and Nox T3 collected during nighttime sleep (1 night)
  Comparisons of sleep TST between Fitbit and Nox T3
Fitbit Sense 2 vs. Nox T3 for sleep efficiency (%) | Fitbit and Nox T3 collected during nighttime sleep (1 night)
  Comparisons of SE between Fitbit and Nox T3
Fitbit Sense 2 vs. Nox T3 for sleep stages (%, min) | Fitbit and Nox T3 collected during nighttime sleep (1 night)
  Comparisons of sleep stages (NREM - stage 1-3, REM) between Fitbit and Nox T3
Fitbit Sense 2 vs. Nox T3 for wake after sleep onset (min) | Fitbit and Nox T3 collected during nighttime sleep (1 night)
  Comparisons of WASO between Fitbit and Nox T3
Fitbit Sense 2 vs. Nox T3 for time of sleep onset and wake time | Fitbit and Nox T3 collected during nighttime sleep (1 night)
  Comparisons of sleep onset time and wake time between Fitbit and Nox T3

SECONDARY OUTCOMES:
Fitbit Sense 2 vs. Sleep Diary for total sleep time (min) | Collected during nighttime sleep (1 night)
  Comparisons of total sleep time between Fitbit and self-reported sleep diary.
Fitbit Sense 2 vs. Sleep Diary for sleep efficiency (%) | Collected during nighttime sleep (1 night)
  Comparisons of sleep efficiency between Fitbit and self-reported sleep diary.
Fitbit Sense 2 vs. Sleep Diary for time of sleep schedule | Collected during nighttime sleep (1 night)
  Comparisons of time of sleep between Fitbit and self-reported sleep diary.
Fitbit Sense 2 vs. Sleep Diary for wake after sleep onset (min) | Collected during nighttime sleep (1 night)
  Comparisons of WASO between Fitbit and self-reported sleep diary.
Subgroup analysis based on gender | Collected at study baseline
  Gender-based subgroup analysis of outcomes
Subgroup analysis based on comorbidities | Collected at study baseline
  Descriptive data on participant comorbidities (e.g., presence of mobility limiting conditions, etc; yes/no) or subgroup analysis by comorbidities
Subgroup analysis based on use of walking aids | Collected at study baseline
  Subgroup analysis by walking aid usage or descriptive data on walking aid use among participants (e.g., yes vs. no)

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This study requested sharing of IPD in the ethics application.